CLINICAL TRIAL: NCT04382287
Title: Comparison of Clinical Efficacy of MI PASTE Plus® and REMIN PRO® for the Remineralisation of Enamel White Spot Lesions in Primary Teeth
Brief Title: Comparison of Remineralisation Efficacy of MI PASTE Plus® and REMIN PRO® for White Spot Lesions in Primary Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Responsible Party: Principal Investigator, José Arturo Garrocho Rangel, Ph.D., Universidad Autonoma de San Luis Potosí
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JRangel
Record Dates: First submitted 2020-05-05; First posted 2020-05-11 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: White Spot Lesion
Keywords: Primary teeth; Enamel; Remineralisation

STUDY DESIGN:
Intervention Model Description: A randomised double-blind clinical trial, with three parallel study groups (two experimental and one control), whose participants were randomly assigned to one of te three groups.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The three provided pastes had a similar physical appearance
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- REMIN paste (Experimental): The child's parents or caregivers were provided with printed instructions for applying the paste at home. The indicated procedure was as follows: application of the remineralisation agent was limited to the tooth's vestibular surface twice a day, after conventional toothbrushing (both in the morning and at night). The maximal amount of paste to be applied was equal to a pea-sized portion (one finger) per surface. The paste was applied using the parent or caregiver's finger across the WSL surface. After the application of the paste, patients were asked to avoid eating or drinking anything for the next hour.
  Interventions: Procedure: Remin Pro® and MI Paste Plus®
- MI PASTE PLUS (Experimental): The child's parents or caregivers were provided with printed instructions for applying the paste at home. The indicated procedure was as follows: application of the remineralisation agent was limited to the tooth's vestibular surface twice a day, after conventional toothbrushing (both in the morning and at night). The maximal amount of paste to be applied was equal to a pea-sized portion (one finger) per surface. The paste was applied using the parent or caregiver's finger across the WSL surface. After the application of the paste, patients were asked to avoid eating or drinking anything for the next hour.
  Interventions: Procedure: Remin Pro® and MI Paste Plus®
- COLGATE Total (Active Comparator): The child's parents or caregivers were provided with printed instructions for applying the paste at home. The indicated procedure was as follows: application of the remineralisation agent was limited to the tooth's vestibular surface twice a day, after conventional toothbrushing (both in the morning and at night). The maximal amount of paste to be applied was equal to a pea-sized portion (one finger) per surface. The paste was applied using the parent or caregiver's finger across the WSL surface. After the application of the paste, patients were asked to avoid eating or drinking anything for the next hour.
  Interventions: Procedure: Remin Pro® and MI Paste Plus®

INTERVENTIONS:
Procedure: Remin Pro® and MI Paste Plus® — Te toothastes were applied at home twice a day over the six anterior upper primary teeth

SUMMARY:
The present study aimed to compare the remineralisation capacity of white spot enamel lesions between two commercially available tooth pastes (Remin Pro and MI PASTE PLUS), applied at home twice a day on the anterior upper primary teeth by the patient and parents.

DETAILED DESCRIPTION:
Objective: To evaluate and compare the clinical efficacy of Remin Pro® and MI Paste Plus® for the remineralisation of white spot lesions (WSL) on the enamel of primary teeth.

Methods: The selected design for this study was a randomised double-blind clinical trial based on CONSORT guidelines. Patients with at least one upper anterior primary tooth with a WSL on the enamel surface, with units of fluorescence (UF) ranged from 11-20 (evaluated with DIAGNOdent) were included in the study. Patients were randomly assigned to receive either the twice-daily at-home topical application of Remin Pro® or MI Paste Plus® (both as experimental pastes) or Colgate Total® (as control paste). The degree of remineralisation was quantified by the change in the number of UF from the baseline evaluation and at days 10 and 21. The difference between groups was statistically evaluated using ANCOVA and ANOVA techniques.

ELIGIBILITY:
Inclusion Criteria:

* Young paediatric patients with at least one upper anterior primary tooth exhibiting one or several WSL on the smooth enamel surface.
* Attending the Paediatric Dentistry Postgraduate Program's Clinic
* Enamel lesions with units of fluorescence (UF) ranging from 11-20 as determined by DIAGNOdent
* Signed Informed Consent

Exclusion Criteria:

* History of hypersensitivity to any of the compounds of the pastes
* Enamel hypoplasia
* Compromising systemic diseases

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 123 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Enamel remineralisation degree | 10 days
  The remineralisation degree was quantified by the change in UF from the baseline (0 day) up to day 10 of twice-daily applications, by evaluation on the 10th day.
Enamel remineralisation degree | 21 days
  The remineralisation degree was quantified by the change in UF from the 10th day up to the 21st day, after twice-daily applications

CONTACTS AND LOCATIONS:
Overall Officials: Amaury Pozos-Guillén, PhD, Study Director — San Luis Potosi University
Locations (1):
- Faculty of Dentistry, Universidad Autónoma de san Luis Potosi, San Luis Potosí City, Mexico

IPD SHARING:
Plan to Share IPD: No